CLINICAL TRIAL: NCT05695040
Title: Evaluation of the Implementation of a Diet Workshop on the 15th Postoperative Day Following Bariatric Surgery on the Protein Intake of the Patient
Brief Title: Evaluation of the Implementation of a Diet Workshop on the 15th Postoperative Day Following Bariatric Surgery
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2020 RODA; 2020-A03239-30 (Other: 2020-A03239-30)
Record Dates: First submitted 2023-01-13; First posted 2023-01-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary workshop conducted on the 15th postoperative day (Experimental)
  Interventions: Behavioral: dietary workshop "proteins"
- Standard care (No Intervention)

INTERVENTIONS:
Behavioral: dietary workshop "proteins" — The workshop will have 2 objectives:
  * Information of the importance of protein after bariatric surgery and the different sources of protein in the diet.
  * Manipulation of a tool in the form of a real size and shape stomach (before and after surgery) that patients will be able to fill and manipulate in order to visualize the quantities needed to achieve the sensation of satiety.
  Arms: dietary workshop conducted on the 15th postoperative day

SUMMARY:
The objective of the study was to improve protein intake after the implementation of a dietary workshop performed on the 15th postoperative day following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 18 years of age
* Scheduled for bariatric surgery such as sleeve gastrectomy or bypass surgery.
* Able to give informed consent to participate in the research.
* Enrolled in a Social Security system.

Exclusion Criteria:

* Inability to travel to participate in the workshop.
* Patients with a diet excluding animal proteins (vegetarians, vegans).
* Pregnant and lactating women.
* Inability to comply with protocol recommendations.
* Incapacitated patients.
* Major deprived of liberty
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Protein intake | 1, 3, 6, and 12 months
  Different measurements of protein intake will be performed at 1, 3, 6, and 12 months in order to observe an improvement in the kinetics of protein intake, the objective being to increase protein intake in the year following surgery and not only at a specific time.

SECONDARY OUTCOMES:
Patient's biometric parameters. Muscle function The patient's muscle mass. Undernutrition Nitrogen balance (ancillary ) Medico-economic evaluation | 3, 6 and 12 months
  -Evaluate the effect of the diet workshop at 3, 6 and 12 months on: The patient's biometric parameters. Muscle function The patient's muscle mass. Undernutrition Nitrogen balance (ancillary ) Medico-economic evaluation
Qualitative evaluation of the workshop at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica RODA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France